CLINICAL TRIAL: NCT04132050
Title: A Phase III Study in Patients With Chronic Idiopathic Thrombocytopenic Purpura in R788
Brief Title: A Clinical Study in Patients With Chronic Idiopathic Thrombocytopenic Purpura in R788
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R788-1301
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2023-12

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R788 (Experimental): Patients are administered R788 for 24 weeks (double-blind period), followed by R788 for up to 52 weeks (open-label period). Patients who have completed open-label period and meet the criteria are eligible to continue R788 treatment over a 3 year period (extension - period).
  Interventions: Drug: R788
- Placebo (Placebo Comparator): Patients are administered Placebo for 24 weeks (double-blind period), followed by R788 for up to 28 weeks (open-label period). Patients who have completed open-label period and meet the criteria are eligible to continue R788 treatment over a 3 year period (extension - period).
  Interventions: Drug: R788; Drug: Placebo

INTERVENTIONS:
Drug: R788 — Oral administration
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy, safety and pharmacokinetics of R788 compared with placebo, and to investigate the safety and efficacy of long term dosing of R788 in patients with chronic idiopathic thrombocytopenic purpura.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients
* Patients diagnosed with idiopathic thrombocytopenic purpura at least 6 months before acquisition of consent
* Patients with a platelet count averages <30000/μL during screening period. Each platelet count should not exceed 35000/μL.
* Patients who have used and failed or who were intolerant at least 1 typical regimen for the treatment of ITP before informed consent (with or without splenectomy)

Exclusion Criteria:

* Patients with thrombocytopenia associated with other disease
* Patients with autoimmune hemolytic anemia
* Patients with poorly controlled hypertension
* Patients with a history or active coagulopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2023-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-two subjects were screened. Of these, 34 subjects considered eligible for the study were randomized to receive the investigational products. The number of subjects in Period I were 22 in the R788 group and 12 in the placebo group. The number of subjects who completed Period I was 10 in the R788 group and 4 in the placebo group.
Groups:
- R788 Group: R788 will be administered orally for 24 weeks in the Period I.
- Placebo Group: R788 placebo will be administered orally for 24 weeks in the Period I.
Period: Period I (Double-blind Period)
Arm/Group | R788 Group | Placebo Group
Started | 22 | 12
Completed | 10 | 4
Not Completed | 12 | 8
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 9 | 8
Period: R788 Treatment Period
Arm/Group | R788 Group | Placebo Group
Started (R788 was administered to 33 subjects throughout the study. Of these, 22 subjects completed the study and 11 subjects discontinued the study.) | 33 (Subjects in the R788 group of double-blind period will be administered R788 for 24 weeks (double-blind period), followed by R788 for up to 52 weeks (open-label period).Subjects in the placebo group of double-blind period will be administered R788 fo 28 weeks (open-label period). Subjects who have completed open-label period and meet the criteria are eligible to continue R788 treatment over a 3 year period (extension-period).) | 0
Completed | 22 | 0
Not Completed | 11 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Lack of Efficacy | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R788 Group | Placebo Group | Total
Number analyzed (Participants) | 22 | 12 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 7 | 19
  >=65 years | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (15.4) | 60.8 (15.4) | 60.0 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 8 | 26
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 12 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 12 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 22 | 12 | 34
Baseline platelet count [Median (Full Range); unit: cells/μL] | 19000 [3000 to 28000] | 18000 [1000 to 27000] | 18000 [1000 to 28000]
Time since ITP diagnosis [Median (Full Range); unit: years] | 12 [1 to 41] | 12 [1 to 38] | 12 [1 to 41]
History of splenectomy [Count of Participants; unit: Participants] | 5 | 2 | 7
Line of Therapy [Count of Participants; unit: Participants]
  2 | 10 | 4 | 14
  ≥3 | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Achievement Rate of Stable Platelet Response
Description: The percentage of subjects who achieved stable platelet response (defined as a platelet count of ≥50000/μL at 4 or more of the 6 visits from Weeks 14 to 24)
Time Frame: 24 weeks (Period I)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | R788 Group | Placebo Group
Number analyzed (Participants) | 22 | 12
Percentage of participants | 36.4 [17.2 to 59.3] | 0.0 [0.0 to 26.5]
Statistical Analysis 1: Comparison: R788 Group vs Placebo Group; Test type: Superiority; p = 0.030, Fisher Exact; Difference in Percent of Participants = 36.4, 95% CI 2-sided [3.1 to 59.3] — The difference in the achievement rate of "Stable platelet response" (= platelet count of ≥ 50000/μL at 4 or more of the 6 visits from Weeks 14 to 24) between two groups and its two-sided 95% CI were calculated

2. Other Pre Specified Outcome: Duration of Platelet Response
Description: Period from the first measurement day on which a platelet count of ≥50000/μL for at least 28 consecutive days was achieved to the first measurement day on which platelet count fell below 50000/μL for at least 28 consecutive days
Time Frame: R788 treatment period (maximum duration of exposure was 1184 days)
Measure: Median (Full Range); unit: days
Groups:
- R788 Group: Subjects in the R788 group of double-blind period will be administered R788 for 24 weeks (double-blind period), followed by R788 for up to 52 weeks (open-label period).Subjects in the placebo group of double-blind period will be administered R788 fo 28 weeks (open-label period). Subjects who have completed open-label period and meet the criteria are eligible to continue R788 treatment over a 3 year period (extension-period).
Arm/Group | R788 Group
Number analyzed (Participants) | 33
days | 392 [106 to 946]

ADVERSE EVENTS:
Time Frame: - Period I: 24 weeks - R788 treatment period: Period I (24 weeks) + Period II (28 weeks) + Period III (Period III and the period of post-marketing clinical study: Maximum 845 days)
Description: Although the time frames are different, the AEs observed in the R788 group and Placebo groups in Period I (double-blind) and the AEs collected from all subjects who received R788 throughout the R788 Treatment Period (double-blind + open-label (including post-marketing study)) are listed in the same table.
Groups:
- R788 Group (Period I): R788 will be administered orally for 24 weeks. On Day 1, 100 mg of the investigational product will be administered. The dose of 100 mg of the study drug will be administered and this must be the only administration of the study drug on Day 1, irrespective of the time of administration. The investigational product will be administered twice daily beginning on the next day (=100 mg bid). If the platelet count at Week 4 or later is below 50000/μL and the investigational product has been well tolerated, the dose of investigational product will be increased from 100 mg bid to 150 mg bid at the discretion of the investigator. The dose during Period I will be adjusted in accordance with the platelet count and tolerance to the investigational product.
- Placebe Group (Period I): R788 placebo will be administered orally for 24 weeks. On Day 1, 100 mg of the investigational product will be administered. The dose of 100 mg of the study drug will be administered and this must be the only administration of the study drug on Day 1, irrespective of the time of administration. The investigational product will be administered twice daily beginning on the next day (=100 mg bid). If the platelet count at Week 4 or later is below 50000/μL and the investigational product has been well tolerated, the dose of investigational product will be increased from 100 mg bid to 150 mg bid at the discretion of the investigator. The dose during Period I will be adjusted in accordance with the platelet count and tolerance to the investigational product.
- R788 Group (R788 Treatment Period): * Period I: R788 will be administered orally for 24 weeks as detailed left.
  * Period II: R788 will be administered orally for 28 weeks.
  * Period III: R788 will be administered orally until market authorization of R788 in Japan.
  * Period of post-marketing study: R788 will be administered orally shall be from the date of market authorization of R788 to the date of first scheduled visit after the day on which R788 becomes available for use as a marketed product to the subject.
  The dose of R788 is adjusted up or down depending on the platelet count within the range of 100 mg qd, 100 mg bid, 150 mg qd, and 150 mg bid.
Arm/Group | R788 Group (Period I) | Placebe Group (Period I) | R788 Group (R788 Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/12 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/22 | 1/12 | 8/33
Other Adverse Events (participants affected / at risk) | 15/22 | 7/12 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R788 Group (Period I) (N=22) | Placebe Group (Period I) (N=12) | R788 Group (R788 Treatment Period) (N=33)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R788 Group (Period I) (N=22) | Placebe Group (Period I) (N=12) | R788 Group (R788 Treatment Period) (N=33)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 6 (6)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (5)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 7 (8) | 1 (1) | 11 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (17) | 0 (0) | 13 (26)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (3) | 0 (0) | 2 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 2 (3)
Blood pressure increased (Investigations) | 1 (2) | 0 (0) | 2 (3)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 4 (5)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0) | 3 (4)
Procedural haemorrhage (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT04132050/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT04132050/SAP_001.pdf